CLINICAL TRIAL: NCT06617832
Title: Trial Designs for Evaluating Migraine Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: UAarhus_Acute migraine
Record Dates: First submitted 2024-09-20; First posted 2024-10-01 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-09

CONDITIONS: Migraine with Aura; Migraine Without Aura; Headache, Migraine
Keywords: Headache; Episodic migraine; Randomized controlled trial; Balanced placebo design; Treatment effects; Adverse events
MeSH Terms: conditions — Migraine with Aura; Migraine without Aura; Migraine Disorders; Headache

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized controlled cross-over design where patients receive 1) sumatriptan or 2) placebo and are told that they receive a) sumatriptan or placebo, b) sumatriptan, or c) placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active group (Active Comparator): Active drug
  Interventions: Drug: Active drug for acute migraine treatment
- Placebo group (Placebo Comparator): Inactive placebo
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Active drug for acute migraine treatment — Standard dose of Sumatriptan 100 mg, which is used as an acute treatment for episodic migraine
  Arms: Active group
Drug: Placebo Oral Tablet — Inactive placebo pill (100 mg) looking like the active drug
  Arms: Placebo group

SUMMARY:
The study aims to estimate treatment effects in randomized controlled trials (RCT) and a balanced placebo design (BPD) to specify how contextual and psychological factors interact in acute migraine treatment and influence adverse event occurrence. Using a clinical within-subjects design, patients with episodic migraine will receive six treatment conditions in a randomized order.

DETAILED DESCRIPTION:
The existing paradigm for testing the effect of treatments is the double-blind RCT comparing an active drug to an inactive placebo. This comparison is done in order to control for contextual and psychological factors such as the patients' treatment expectations - a key factor in placebo responses. However, recent study results have indicated that some assumptions underlying the RCT may be incorrect and may lower the assay sensitivity and miscalculate the actual drug response. The so-called balanced placebo design targets the shortcomings of the RCT by balancing the information given to the patients (correct or false) with the actual treatment administered (active treatment or placebo). In this project, the aim is to examine if the magnitude of the drug effect differs when estimated based on the RCT design and when based on BPD, conditioning on the information provided to the recipient. Additionally, it will also be tested if active drug response and the placebo response interact in acute migraine treatment.

Patients suffering from episodic migraine will go through six treatment conditions in randomized order. They will receive acute migraine treatment (a sumatriptan pill) or inactive treatment (a placebo pill) in the event of a developing migraine attack. Using a clinical within-subjects design, the patients receive 1) sumatriptan or 2) placebo and are told that they receive a) sumatriptan or placebo, b) sumatriptan , or c) placebo. All treatments and accompanying treatment descriptions will be administered at home.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18-65 years)
2. ≥ 1-year history of migraine with or without aura according to the International Classification of Headache Disorders (ICHD-3) diagnostic criteria
3. Known episodic migraine (≥ 1 and < 15 headache days with features of migraine on at least 2-8 days per month for > 3 months) with and without aura and diagnosed before age 50
4. Previous or active use of triptans as acute treatment for migraine
5. Ability to speak and read Danish

Exclusion Criteria:

1. Chronic migraine or history of chronic migraine in the last 12 months
2. Other concomitant primary headache types except for infrequent tension-type headache
3. Secondary headache disorders including medication overuse headache
4. Severe psychiatric, vascular or liver diseases
5. Opioid or barbiturate use in the month preceding screening
6. Current use of preventive migraine treatment (i.e., onabotulinum toxin A, and/or Calcitonin gene-related peptide (CGRP) monoclonal antibodies) (however, stable medical treatment with other migraine prophylactic agents is permitted, e.g. antidepressant, calcium channel blockers, beta blockers and antiepileptic drugs, 4 weeks prior to baseline until the completion of participation in the study)
7. Contraindications or inability to tolerate triptans
8. Current substance use disorder
9. Implanted metallic or electronic device in the head
10. Cardiac pacemaker or implanted or wearable defibrillator
11. Use of illegal psychotropic drugs less than a week before participation in the study; regarding cannabis: less than four weeks before participation in the study
12. Current pregnancy or planned pregnancy (confirmed by pregnancy test and by use of safe contraception as defined by the Danish Medicines Agency) and lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Headache intensity | 2 hours from each treatment administration
  Headache intensity rated on a 11-point Numerical Rating Scale (0=no pain; 10=worst imaginable pain) 2 hours after each treatment condition.
Adverse events | 2 hours from each treatment administration
  Occurrence of adverse events in each treatment condition recorded by the presence of adverse events ascribed to the treatment, measured by free recall and by prompting.

SECONDARY OUTCOMES:
Positive and negative affect (PANAS) | Before and 2 hours after each treatment administration
  PANAS will be used to measure positive and negative emotions or feelings in the present moment. Positive affectivity refers to positive emotions and expressions. Negative affectivity, on the other hand, refers to negative emotions and expressions. This scale consists of words that describe different emotions and is scored on a likert scale ranging from 1 to 5 (1= Very slightly or Not at all, 2=little, 3=moderately, 4=quite a bit and 5 =extremely).
Functional disability scale | Before and 2 hours after each treatment administration
  Functional disability due to migraine will be measured on a 4-point scale (0= no disability (i.e., able to function normally); 1=mild disability (i.e., able to perform all activities of daily living but with some difficulty); 2=moderate disability (i.e., unable to perform certain activities of daily living); 3=severe disability (i.e., unable to perform most to all activities of daily living or requiring bed rest)
Rescue medication | 2 hours from each treatment administration
  Use of rescue medication for episodic migraine (type of rescue medications and time of administration) will be noted
Pain Freedom | 2 hours from each treatment administration
  Freedom from pain will be measured as yes/no at 2 hours after each treatment condition
Absence of the most bothersome symptom | 2 hours from each treatment administration
  Absence of the most bothersome migraine-associated symptoms such as nausea, vomiting, photophobia, and phonophobia. The participants are asked to answer the question by answering yes or no.
Intensity of experienced adverse events | 2 hours (from each treatment administration)
  Intensity of the experienced adverse events will be measured on a 11-point Numerical Rating Scale (e.g., "To what extent have you been feeling fatigue/dizziness?"; 0=not at all; 10=worst imaginable)

OTHER OUTCOMES:
Expectations | Before administration of each treatment condition
  Expectations regarding the treatment effect and the occurrence of adverse events will be measured on a 11-point Numerical Rating Scale (e.g., "How likely do you think it is that you will experience adverse events from the treatment?"; 0=not at all; 10=extremely likely). This parameter is measured as a predictor rather than an outcome measure

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Dept. of Psychology and Behavioural Sciences, Aarhus C
  - Department of Clinical Medicine, Aarhus University Hospital, Aarhus N

IPD SHARING:
Plan to Share IPD: No